CLINICAL TRIAL: NCT06583291
Title: A Single Center, Open-label Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Allogeneic Dopaminergic Neural Precursor Cell(iDAP) Injection in the Treatment of Parkinson's Disease
Brief Title: iDAP Injection in the Treatment of Parkinson's Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCR201-1001
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): MRI-guided bilateral stereotactic cell implantation
  Interventions: Drug: Allogeneic dopaminergic neural precursor cell(iDAP)
- High dose (Experimental): MRI-guided bilateral stereotactic cell implantation
  Interventions: Drug: Allogeneic dopaminergic neural precursor cell(iDAP)

INTERVENTIONS:
Drug: Allogeneic dopaminergic neural precursor cell(iDAP) — Bilateral implantation

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and preliminary efficacy that iDAP has on Parkinson's disease (PD) patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease in the middle-aged and elderly. It is the "third killer" of the middle-aged and elderly after tumors and cardiovascular and cerebrovascular diseases. Its main clinical manifestations are resting tremor, reduced voluntary movement, muscle rigidity, postural reflex impairment, and autonomic dysfunction, which seriously affect patients' work ability and quality of life. It is estimated that nearly 100,000 people in China become new Parkinson's patients every year. Experts from the World Health Organization predict that the number of Parkinson's patients in China will reach 5 million in 2030, which will be more than half of the world's total. As the disease progresses, the symptoms of Parkinson's patients will become increasingly severe. The high prevalence and high disability rate of Parkinson's disease bring heavy burdens to individuals, families, and society.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 45 and 75 years;
* Diagnosed to be Parkinson's disease patients according to MDS Parkinson's disease diagnostic criteria;
* Disease history 4-20 years;
* Hoehn and Yahr Stage 2-4;
* Stable dose of dopamine for more than 3 months;
* Improvement of MDS-UPDRS part III;

Exclusion Criteria:

* Patients who have previously undergone brain surgery;
* Past use of stem cell therapy or participation in stem cell clinical research;
* Cognitive impairment;
* History of mental disorders;
* Patients with other serious systemic diseases;
* Past or current metastatic malignant tumors.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | Within 24 months post-transplantation
  Safety and tolerability

SECONDARY OUTCOMES:
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part III, in comparison with baseline values. | Within 24 months post-transplantation
  Minimum score: 0; Maximum score: 132; Higher scores mean a worse outcome.
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part I,II,IV, in comparison with baseline values. | Within 24 months post-transplantation
  Higher scores mean a worse outcome.
Assessment of changes in Hoehn & Yahr scale in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in Parkinson disease.
Assessment of changes in Mini-mental State Examination (MMSE), Hamilton Depression Scale (HAMD)-17 and Hamilton Anxiety Scale (HAMA)-14 in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in mental state.
Assessment of changes in Activity of Daily Living Scale (ADL) in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in activity of daily living.
Brain network connectivity patterns as demonstrated on positron emission tomography(PET) compared with baseline in the 'off' state. | Within 24 months post-transplantation
  Evidence of cell survival
Brain DAT intake index as demonstrated on PET dopamine transporter(DAT) compared with baseline in the 'off' state. | Within 24 months post-transplantation
  Evidence of cell survival
Patient L-dopa equivalent dose compared with baseline. | Within 24 months post-transplantation
  Measure of dopaminergic drug dose.

IPD SHARING:
Plan to Share IPD: No